CLINICAL TRIAL: NCT04632290
Title: Brain-controlled Spinal Cord Stimulation in Patients With Spinal Cord Injury
Acronym: STIMO-BSI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Prof., Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STIMO-BSI
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants receive the same intervention.
  Interventions: Device: STIMO-BSI system implantation; Device: ARC-BSI Lumbar System

INTERVENTIONS:
Device: STIMO-BSI system implantation — Participants are implanted bilaterally with epidural electrocorticography devices. The decoded motor intentions are driving the implanted spinal cord stimulation system. Brain-controlled spinal cord stimulation is used for training and rehabilitation to recover voluntary movements.
Device: ARC-BSI Lumbar System — ARC-BSI Lumbar System for participants entering the optional extension with system upgrade: replacement of the neurostimulator, and upgrade of the WIMAGINE system and STIMO system wearable devices.

SUMMARY:
In a current first-in-human study, called Stimulation Movement Overground (STIMO, NCT02936453), Epidural Electrical Stimulation (EES) of the spinal cord is applied to enable individuals with chronic severe spinal cord injury (SCI) to complete intensive locomotor neurorehabilitation training. In this clinical feasibility study, it was demonstrated that EES results in an immediate enhancement of walking function, and that when applied repeatedly as part of a neurorehabilitation program, EES can improve leg motor control and trigger neurological recovery in individuals with severe SCI to a certain extent (Wagner et al. 2018).

Preclinical studies showed that linking brain activity to the onset and modulation of spinal cord stimulation protocols not only improves the usability of the stimulation, but also augments neurological recovery. Indeed, rats rapidly learned to modulate their cortical activity in order to adjust the amplitude of spinal cord stimulation protocols. This brain-spine interface allowed them to increase the amplitude of the movement of their otherwise paralyzed legs to climb up a staircase (Bonizzato et al. 2018). Moreover, gait rehabilitation enabled by this brain-spine interface (BSI) augmented plasticity and neurological recovery. When EES was correlated with cortical neuron activity during training, rats showed better recovery than when training was only supported by continuous stimulation (Bonizzato et al. 2018). This concept of brain spine-interface was validated in non-human primates (Capogrosso et al. 2016).

Clinatec (Grenoble, France) has developed a fully implantable electrocorticogram (ECoG) recording device with a 64-channel epidural electrode array capable of recording electrical signals from the motor cortex for an extended period of time and with a high signal to noise ratio the electrical signals from the motor cortex. This ECoG-based system allowed tetraplegic patients to control an exoskeleton (ClinicalTrials.gov, NCT02550522) with up to 8 degrees of freedom for the upper limb control (Benabid et al. 2019). This device was implanted in 2 individuals so far; one of them has been using this system both at the hospital and at home for more than 3 years.

We hypothesize that ECoG-controlled EES in individuals with SCI will establish a direct bridge between the patient's motor intention and the spinal cord below the lesion, which will not only improve or restore voluntary control of leg movements, but will also boost neuroplasticity and neurological recovery when combined with neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Having completed the main phase of the STIMO study (NCT02936453).
* SCI graded as American Spinal Injury Association Impairment Scale (AIS) A, B, C & D
* Level of lesion: T10 and above, based on AIS level determination by the PI, with preservation of conus function
* The intact distance between the cone and the lesion must be at least 60 mm.
* Focal spinal cord disorder caused by either trauma or epidural, subdural or intramedullary bleeding
* Minimum 12 months post-injury
* Completed in-patient rehabilitation program
* Stable medical, physical and psychological condition as considered by Investigators
* Able to understand and interact with the study team in French or English
* Adequate care-giver support and access to appropriate medical care in patient's home community
* Must agree to comply in good faith with all conditions of the study and to attend all required study training and visit
* Must provide and sign the Informed Consent prior to any study related procedures

Exclusion Criteria:

* Limitation of walking function based on accompanying (CNS) disorders (systemic malignant disorders, cardiovascular disorders restricting physical training, peripheral nerve disorders)
* History of severe autonomic dysreflexia
* Brain damage
* Epilepsy
* Spinal stenosis
* Use of an intrathecal Baclofen pump.
* Any active implanted cardiac device such as pacemaker or defibrillator.
* Any indication that would require diathermy.
* Any indication that would require MRI.
* Increased risk for defibrillation.
* Severe joint contractures disabling or restricting lower limb movements.
* Haematological disorders with increased risk for surgical interventions (increased risk of haemorrhagic events).
* Congenital or acquired lower limb abnormalities (affection of joints and bone).
* Women who are pregnant (pregnancy test obligatory for women of childbearing potential) or breast feeding or not willing to take contraception.
* Known or suspected non-compliance, drug or alcohol abuse.
* Spinal cord lesion due to either a neurodegenerative disease or a tumor.
* Gastrointestinal ulcers in the last five years
* Known or suspected eye disorders or diseases
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Any other anatomic or co-morbid conditions that, in the investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow-up requirements, or impact the scientific soundness of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-07-04 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Safety Measure | Through study completion, an average of 1 year
  Number of Adverse Events possibly, probably or causally related to the procedure or device.
Safety Measure | Through study completion, an average of 1 year
  Number of device deficiencies

SECONDARY OUTCOMES:
WISCI II score | 1 week before implantation, 8 weeks and 19 weeks after implantation
  From 0 to 20, higher scores mean a better outcome
10mWT | 1 week before implantation, 8 weeks and 19 weeks after implantation
Weight bearing capacity | 1 week before implantation, 8 weeks and 19 weeks after implantation
SCIM III score | 1 week before implantation, 8 weeks and 19 weeks after implantation
  From 0 to 100, higher scores mean a better outcome
6minWT | 1 week before implantation, 8 weeks and 19 weeks after implantation
Time Up and Go | 1 week before implantation, 8 weeks and 19 weeks after implantation
Maximum Voluntary Contraction | 1 week before implantation, 8 weeks and 19 weeks after implantation
ASIA score | 1 week before implantation, 8 weeks and 19 weeks after implantation
  From 0 to 100, higher scores mean a better outcome
Modified Ashworth Scale | 1 week before implantation, 8 weeks and 19 weeks after implantation
  From 0 to 4, higher scores mean a worst outcome
Berg Balance Scale | 1 week before implantation, 8 weeks and 19 weeks after implantation
  From 0 to 56, higher scores mean a better outcome
Gait Analysis | 1 week before implantation, 8 weeks and 19 weeks after implantation
  Average step height, step length, amplitude of EMG activity during walking
WHOQOL-BREF | 1 week before implantation, 8 weeks and 19 weeks after implantation
  From 0 to 100, higher scores mean a better outcome
BCI performance measures | 8 weeks and 19 weeks after implantation
  Decoding accuracy from 0-100% higher numbers mean a better outome
Upper Limb Neurobiomechanics | 8 weeks and 19 weeks after implantation
  Average range of movement, amplitude of EMG activity during upper limb movements
ECoG signal stability | 8 weeks and 19 weeks after implantation
  Power density spectrum of the ECoG signal over each electrode
SSEP | 8 weeks and 19 weeks after implantation
  Amplitude and latency of the cortically evoked potentials

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Capogrosso M, Milekovic T, Borton D, Wagner F, Moraud EM, Mignardot JB, Buse N, Gandar J, Barraud Q, Xing D, Rey E, Duis S, Jianzhong Y, Ko WK, Li Q, Detemple P, Denison T, Micera S, Bezard E, Bloch J, Courtine G. A brain-spine interface alleviating gait deficits after spinal cord injury in primates. Nature. 2016 Nov 10;539(7628):284-288. doi: 10.1038/nature20118. PMID 27830790
- [Background] Benabid AL, Costecalde T, Eliseyev A, Charvet G, Verney A, Karakas S, Foerster M, Lambert A, Moriniere B, Abroug N, Schaeffer MC, Moly A, Sauter-Starace F, Ratel D, Moro C, Torres-Martinez N, Langar L, Oddoux M, Polosan M, Pezzani S, Auboiroux V, Aksenova T, Mestais C, Chabardes S. An exoskeleton controlled by an epidural wireless brain-machine interface in a tetraplegic patient: a proof-of-concept demonstration. Lancet Neurol. 2019 Dec;18(12):1112-1122. doi: 10.1016/S1474-4422(19)30321-7. Epub 2019 Oct 3. PMID 31587955
- [Background] Bonizzato M, Pidpruzhnykova G, DiGiovanna J, Shkorbatova P, Pavlova N, Micera S, Courtine G. Brain-controlled modulation of spinal circuits improves recovery from spinal cord injury. Nat Commun. 2018 Aug 1;9(1):3015. doi: 10.1038/s41467-018-05282-6. PMID 30068906